CLINICAL TRIAL: NCT02385877
Title: Clinical Translation of 18F-Labeled Hydroxyphenethylguanidines for Quantification of Regional Cardiac Sympathetic Nerve Density With PET
Brief Title: Clinical Translation of 18F-Labeled Hydroxyphenethylguanidines
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David M. Raffel, Ph.D., Research Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00088601
Record Dates: First submitted 2015-02-25; First posted 2015-03-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Autonomic Peripheral Nervous System Diseases
MeSH Terms: conditions — Autonomic Nervous System Diseases | interventions — 4-fluoro-3-hydroxyphenethylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Protocol 1: [18F]4F-MHPG (Experimental): Subjects (n = 4) will be injected one time with 6.5 mCi of 4-[18F]fluoro-meta-hydroxyphenethylguanidine ([18F]4F-MHPG) and receive a 90 minute PET scan.
  Interventions: Drug: [18F]4F-MHPG
- Protocol 1: [18F]3F-PHPG (Experimental): Subjects (n = 4) will be injected one time with 6.5 mCi of 3-[18F]fluoro-para-hydroxyphenethylguanidine ([18F]3F-PHPG) and receive a 90 minute PET scan.
  Interventions: Drug: [18F]3F-PHPG
- Protocol 2: Biodistribution Studies (Experimental): Subjects (n = 4) will be injected one time with 6.5 mCi of either [18F]4F-MHPG or [18F]3F-PHPG (whichever is selected based on Protocol 1 studies) and receive four whole-body PET scans, starting at 5 min, 60 min, 150 min and 360 min after tracer injection.
  Interventions: Drug: [18F]4F-MHPG; Drug: [18F]3F-PHPG

INTERVENTIONS:
Drug: [18F]4F-MHPG — IV injection of [18F]4F-MHPG
  Other Names: 4-[18F]fluoro-meta-hydroxyphenethylguanidine
  Arms: Protocol 1: [18F]4F-MHPG; Protocol 2: Biodistribution Studies
Drug: [18F]3F-PHPG — IV injection of [18F]3F-PHPG
  Other Names: 3-[18F]fluoro-para-hydroxyphenethylguanidine
  Arms: Protocol 1: [18F]3F-PHPG; Protocol 2: Biodistribution Studies

SUMMARY:
The purpose of this study is to perform first-in-human PET imaging studies of two new cardiac sympathetic nerve imaging agents, 4-[18F]fluoro-meta-hydroxyphenethylguanidine ([18F]4F-MHPG) and 3-[18F]fluoro-para-hydroxyphenethylguanidine ([18F]3F-PHPG).

DETAILED DESCRIPTION:
In this study, PET imaging studies of two structurally related 18F-hydroxyphenethylguanidines, 4-[18F]fluoro-meta-hydroxyphenethylguanidine ([18F]4F-MHPG) and 3-[18F]fluoro-para-hydroxyphenethylguanidine ([18F]3F-PHPG) will be performed. All studies will be performed in normal healthy volunteers.

PET stands for Positron Emission Tomography which is a type of imaging that uses a radioactive tracer. This is also called a radiotracer which is a compound linked to a radioactive element. Most compounds are short-lived, meaning that the radioactivity breaks down quickly or is excreted from the body.

In the first stage of the study, dynamic PET imaging for 90 min will be done with [18F]4F-MHPG (n = 4) and [18F]3F-PHPG (n = 4).

Data from these studies will assess each radiotracer's imaging properties, pharmacokinetics and metabolic breakdown in plasma. Application of tracer kinetic analysis methods to the kinetics of each tracer in heart and plasma will be studied to see if these methods can provide accurate measurements of regional nerve sympathetic nerve density in the hearts of human subjects. Results from these initial studies will be used to select the lead compound for further studies in patient populations.

In the second stage of the study, whole-body PET imaging studies (n = 4) with the selected lead radiotracer will be performed to acquire data necessary for generating more accurate human radiation absorbed dose estimates.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese (BMI < 30)
* Normal blood pressure
* Normal blood lipid profile
* No history of prior cardiovascular disease
* Not susceptible to claustrophobia
* Ability to lay flat for 90 min

Exclusion Criteria:

* Obesity (BMI > 30)
* Risk factors for heart disease (age > 55y, hypertension, smoking, high blood pressure, high cholesterol levels, diabetes, etc.)
* History of heart disease (heart attack, atrial fibrillation, ventricular tachycardia, exertional angina)
* Currently using certain medications that may interact with cardiac nerves (antidepressants, cold medications, nasal decongestants, monoamine oxidase inhibitors, etc.)
* Claustrophobia
* Inability to lie flat for 90 min
* Pregnant or breast feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Composite measure based on radiotracer tissue uptake ratios (heart-to-lung ratio, heart-to-liver ratio, heart-to-blood ratio) and rates of metabolism in plasma (half-time, in minutes) of [18F]4F-MHPG and [18F]3F-PHPG in healthy subjects. | 3 months
  These data will be used to select the lead radiotracer for further clinical development.

SECONDARY OUTCOMES:
Radiation Dose | 1 year
  Human radiation absorbed dose estimates based on the kinetics of the selected lead radiotracer in various organs, as extracted from whole-body PET scans.
Number of Adverse Events | 30 days
  Number of study participants with adverse events as a measure of safety and tolerability following intravenous administration of [18F]4F-MHPG or [18F]3F-PHPG

CONTACTS AND LOCATIONS:
Overall Officials: David M Raffel, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raffel DM, Jung YW, Koeppe RA, Jang KS, Gu G, Scott PJH, Murthy VL, Rothley J, Frey KA. First-in-Human Studies of [18F] Fluorohydroxyphenethylguanidines. Circ Cardiovasc Imaging. 2018 Dec;11(12):e007965. doi: 10.1161/CIRCIMAGING.118.007965. PMID 30558502